CLINICAL TRIAL: NCT03229304
Title: The Role of Uterine Artery Doppler Measurement to Predict the Amount of Postpartum Hemorrhage in Low Risk Term Pregnancy
Brief Title: Prediction of Postpartum Hemorrhage With Uterine Artery Doppler Measurement
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerem Doga Seckin, ass prof, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 12341
Record Dates: First submitted 2017-07-14; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The aim of the study is to evaluate the uterine artery doppler just before labour in term low risk pregnancies. And to investigate with this measurement if investigators could foreseen the amount of postpartum hemorrhage looking at decreased in the hematocrit values.

ELIGIBILITY:
Inclusion Criteria:

* singleton term pregnancies

Exclusion Criteria:the pregnant women who have

* polyhydramnios
* Large for gestational age fetuses
* multiple pregnancies
* preterm labour
* chorioamnionitis
* history of atonia or postpartum hemorrhage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The pregnant women that is term and have no risk factors for postpartum hemorrhage
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
To measure the uterine artery Pulsatility index in term pregnant women | 6-8 hour before the delivery
  With ultrasonography uterine artery doppler Pulsatility index (cm/s) will be measure
To measure the uterine artery Resistant index (cm/s) in term pregnant women | 6-8 hour before the delivery
  With ultrasonography uterine artery doppler Resistant index will be measure
To measure the uterine artery mean systolic/diastolic volume (cm/s) in term pregnant women | 6-8 hour before the delivery
  With ultrasonography Uterine artery doppler Mean systolic/diastolic volume (cm/s) ) will be measure

CONTACTS AND LOCATIONS:
Locations (1):
- Kerem Doga Seckin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplanoglu M, Karateke A, Un B, Gunsoy L, Baloglu A. Evaluation of uterine artery recanalization and doppler parameters after bilateral uterine artery ligation in women with postpartum hemorrhage. Int J Clin Exp Med. 2015 May 15;8(5):7823-9. eCollection 2015. PMID 26221335
- [Background] Yildirim D, Ozyurek SE, Ekiz A, Eren EC, Hendem DU, Bafali O, Seckin KD. Comparison of active vs. expectant management of the third stage of labor in women with low risk of postpartum hemorrhage: a randomized controlled trial. Ginekol Pol. 2016;87(5):399-404. doi: 10.5603/GP.2016.0015. PMID 27304659